CLINICAL TRIAL: NCT03948425
Title: Cerebral Dynamic Perfusion Study With Spectral CT in Patients Suspected of Stroke
Acronym: AVC_AIGUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AVC AIGUS; 2017/12AVR/209 (Other: CEHF)
Record Dates: First submitted 2018-09-17; First posted 2019-05-14 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke (Experimental): Clinical suspicion of hyperacute stroke (6 hours after onset of symptoms):Intervention 'spectral CT'
  Interventions: Radiation: spectral CT

INTERVENTIONS:
Radiation: spectral CT — Head spectral CT

SUMMARY:
* Generate a dynamic mapping of the distribution of iodine within the cerebral parenchyma in the patient suspected of acute ischemic disorder with the CT spectral scanner.
* Correlate the anomalies of iodine mapping to the other parameters acquired during the classic dynamic infusion phase to define the ischemic area (MTT higher and rCBV normal) versus infarcted zone (MTT higher and rCBV decreased)

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of hyperacute stroke (6 hours after onset of symptoms)
* Age between 50 and 95 years
* Weight: between 65 and 95 kg

Exclusion Criteria:

* Documented or suspected allergy to IV iodinated contrast media
* Renal impairment with creatinine clearance <60 ml / min
* Hemorrhagic lesions or vascular abnormalities demonstrated on CT before contrast injection

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Volume (CBV) | from start of the study procedure (CT scan) through end of study procedure (from 15 minutes to 30 minutes)
  CBV is measured in units of milliliters of blood per 100 g of brain and is defined as the volume of flowing blood for a given volume of brain.
Mean Transit Time (MTT) | rom start of the study procedure (CT scan) through end of study procedure (from 15 minutes to 30 minutes)
  MTT is measured in seconds and defined as the average amount of time it takes blood to transit through the given volume of brain.
Cerebral Blood Flow (CBF) | rom start of the study procedure (CT scan) through end of study procedure (from 15 minutes to 30 minutes)
  CBF is measured in units of milliliters of blood per 100 g of brain tissue per minute and is defined as the volume of flowing blood moving through a given volume of brain in a specific amount of time.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Coche, MD-PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires saint Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duprez T, Vlassenbroek A, Peeters A, Poncelet PA, Levecque E, Austein F, Pahn G, Nae Y, Abdallah S, Coche E. Preliminary experience of CT imaging of the ischaemic brain penumbra through spectral processing of multiphasic CTA datasets. Sci Rep. 2023 Jul 15;13(1):11431. doi: 10.1038/s41598-023-38370-9. PMID 37454162